CLINICAL TRIAL: NCT02411071
Title: Clinical Implications of HIV Low-level Viremia at Times of Highly Active Antiretroviral Treatment Regimens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Essen (Other)
Collaborators: Janssen Medical Affairs (Industry)
Responsible Party: Principal Investigator, Jens Verheyen, PD M.D., University Hospital, Essen
Other Study IDs: 14-6155-BO; TMC114IFD4043 (Other Grant/Funding Number: Janssen-Cilag Medical Affairs EMEA)
Record Dates: First submitted 2015-03-06; First posted 2015-04-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: HIV-infection
Keywords: HIV-1; antiretroviral treatment; low viral load; low-level viremia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Cells and DNA/RNA extracted from whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients starting cART: Patients starting cART. Grouping according to the time needed to reach viral loads below 1000, 500, 400, 200, 50 copies/ml, respectively.
- Patients with cART: Patients with cART. Grouping in patients without and with low-level-viremia (LLV) defined as two consecutive viral loads between 40 copies/ml and 200 copies/ml, 400 copies/ml, 500 copies/ml and 1000 copies/ml, respectively.

SUMMARY:
Retrospective analysis of HIV-1 positive patients treated with antiretroviral therapy in Essen (Germany) from 2004 on. Stored samples from selected patients (n=50) obtained for routine diagnostics will be used to analyze the gag gene, the V3-region of the env gene and immune cells.

DETAILED DESCRIPTION:
The underlying study is a retrospective analysis of HIV-1 positive patients treated with antiretroviral therapy from Essen since 2004. Stored samples obtained for routine diagnostics will be used to analyze the gag gene, the V3-region and immune cells from selected patients. By comparing different groups of patients this study aims to identify clinical implications of low-level viremia (LLV) and persistent viremia (PV) at times of highly active antiretroviral treatment regimens (cART). The objectives of this study is to (1) determine how often LLV and PV occured during cART in Essen in the last 10 years and whether specific patterns can be correlated, (2) whether the evolution of PI drug resistance can be detected earlier in the gag than in the protease gene, (3) what kind of cellular tropism do HIV-1 isolates (RNA and proviral DNA) have at times of LLV, and (4) what kind of immune cells circulate in the blood during LLV and PV and what kind of functional properties do they have. The groups include patients starting cART as well as patients with cART. Furthermore, clinical data of patients are routinely documented and will be combined with results specifically obtained in this study in an anonymized data set. Since this is a retrospective study, there are no specific endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV-1 infection
* Age > 18 years
* Patients treated in Essen in the last 10 years

Exclusion Criteria:

- no antiretroviral therapy / treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A database comprising clinical parameters (viral Ioad, antiretroviral treatment, immunological parameters, HBV/HCV-coinfections and HIV-1 genotypes) of patients treated in Essen in the last 10 years will be set up. These data will be used to compare different groups of patients and will be screened for parameters associated with LLV (defined as two consecutive viral loads between 40 and 1000 copies/ml) or PV (viral loads between above 50 copies/ml 26 weeks after start of ART). Different clinical settings will be distinguished: First patients after the start of first line treatment regimens in the initial phase and second patients after at least 18 months of cART.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Frequencies of low-level viremia (LLV) during ART | In the last 10 years
  Viral loads between 40 and 1000 copies/ml at two consecutive time points preceded by undetectable viral loads
Frequencies of persistant viremia (PV) after start of ART | In the last 10 years
  Viral loads above 50 copies/ml 26 weeks after start of antiretroviral treatment

SECONDARY OUTCOMES:
Patterns associated with LLV or PV | In the last 10 years
  CD4+ cell count, the CD4:CD8 ratio and the number of activated T cells (HLA-DR+), NK-cells (CD3-, CD16+, CD56+) and cytotoxic T-cells (CD3+, CD16+, CCD56+), HBV/HCV Co-Infection status.
Detection of gag mutations | In the last 10 years
HIV tropism during LLV or PV | In the last 10 years
  Determination of the HIV tropism during LLV or PV in a subset of patients
Cellular inflammation markers | In the last 10 years
  Number of Tregs in the peripheral blood. Number of central memory and effector cells.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Verheyen, M.D., Principal Investigator — Institute of Virology, University Duisburg-Essen, University Hospital Essen, Essen, Germany; Stefan Esser, M.D., Principal Investigator — HIV outpatient center, Dept. for Dermatology and Venerolgy, University Duisburg-Essen, University Hospital Essen, Essen, Germany
Locations (1):
- HIV outpatient center, Dept. for Dermatology and Venerolgy, University Duisburg-Essen, University Hospital Essen, Essen, North Rhine-Westphalia, Germany